CLINICAL TRIAL: NCT03718312
Title: Evaluation of the Effectiveness of Ischemic Pre-conditioning on the Morbidity and Mortality of Open Surgery of Thoracoabdominal Aortic Aneurysms.
Acronym: EPICATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/388/HP
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Aortic Aneurysm; Surgery
Keywords: Clamping; pre-conditioning
MeSH Terms: conditions — Aortic Aneurysm | interventions — Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Patients with aortic clamping withpre-conditioning
  Interventions: Procedure: clamping with pre-conditioning (PCl)
- Arm 2 (No Intervention): Patients with aortic clamping without pre-conditioning

INTERVENTIONS:
Procedure: clamping with pre-conditioning (PCl) — PCI procedure: clamping of the supracellular thoracic aorta for 5 minutes followed by a 5-minutes de-clamping period.
  PCI procedure is repeated twice.
  Arms: Arm 1

SUMMARY:
Patients having a planned open surgery of thoracoabdominal aortic aneurysms and enrolled in the study will be randomized the day of the surgery in 2 groups:

* Arm 1 : Patients with aortic clamping with pre-conditioning
* Arm 2 : Patients with aortic clamping without pre-conditioning Patients will be then followed, during 60 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 and <85 years old
2. Patient having a planned surgery for a thoracoabdominal aortic aneurysm by direct approach,
3. Patient with aortic aneurysm requiring supra-visceral aortic clamping and visceral artery reconstruction,
4. Aortic aneurysmal patient with or without distal femoral circulatory assistance,
5. Patient with aortic aneurysm of atheromatous or dissecting etiology,
6. Woman of childbearing potential with effective contraception (estrogen-progestin or intrauterine device or tubal ligation), postmenopausal woman (≥ 12 months of amenorrhea not induced by therapy)
7. Patient who read and understood the newsletter and signed the consent form
8. Patient affiliated with a social security scheme

Exclusion Criteria:

1. Patient with aortic aneurysms requiring supra-visceral aortic clamping but not requiring visceral artery reconstruction (supra-visceral aortic clamping for renal aortic juxtaposition aorta),
2. Patient with thoraco abdominal aortic aneurysms requiring a circulatory arrest (aortic aneurysms affecting the descending thoracic aorta or the aortic arch)
3. Patient requiring emergency aortic surgery
4. Patient under treatment known as interfering with PCI (Nicorandil or oral antidiabetic agents),
5. Pregnant or lactating woman (negative result of baseline blood test)
6. Participation in another interventional study within 28 days before randomization or during this study
7. Person deprived of liberty by an administrative or judicial decision or person subject to a legal measure for the protection of adults,
8. Patient under the protection of justice, patient under guardianship or curatorship.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
occurrence of a pulmonary complication | Before the 48 hours after the beginning surgery
  Need for prolonged invasive ventilation
occurrence of a kidney complication | During the 8 days after surgery
  According to RIFLE criteria
occurrence of a pulmonary complication | During the 8 days after surgery
  Occurrence of a moderate or severe acute respiratory distress syndrome (Berlin definition)
occurrence of a pulmonary complication | During the 48 hours after initial extubation
  Need for a new ventilation (invasive or not)

SECONDARY OUTCOMES:
Pulmonary Morbidity | During the 21 days after surgery
  Need of a new ventilation (invasive or not)
Kidney Morbidity | During the 21 days after surgery
  According to RIFLE criteria
Cardiac Morbidity | During the 48 hours after surgery
  Value of troponin
cell and tissue damage | During the 8 days after surgery
  Value of D Lactate
Death | During 60 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Rouen, Rouen, France

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250
- [Derived] Palmier M, Bubenheim M, Chiche L, Chaufour X, Koskas F, Fadel E, Magnan PE, Ducasse E, Chakfe N, Steinmetz E, Dusseaux MM, Ricco JB, Plissonnier D. Protocol of supra-visceral aortic ischemic preconditioning for open surgical repair of thoracoabdominal aortic aneurysm : The EPICATA study (Evaluation of the Efficacy of Ischemic PreConditioning on morbidity and mortality in open ThoracoAbdominal Aortic surgery). BMC Surg. 2020 Aug 27;20(1):193. doi: 10.1186/s12893-020-00851-3. PMID 32854681